CLINICAL TRIAL: NCT03334058
Title: An Open-label, Non-controlled, Phase II Study to Evaluate the Safety, Pharmacodynamics, Pharmacokinetics, Efficacy and Conditions of Use of ARGX-113 in Patients With Mild to Moderate Pemphigus (Vulgaris and Foliaceus)
Brief Title: A Study to Evaluate the Safety, PD, PK and Efficacy of ARGX-113 in Patients With Pemphigus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARGX-113-1701; 2017-002333-40 (EudraCT Number)
Record Dates: First submitted 2017-10-23; First posted 2017-11-07 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-11

CONDITIONS: Pemphigus Vulgaris; Pemphigus Foliaceus
MeSH Terms: conditions — Pemphigus | interventions — efgartigimod alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ARGX-113 (Experimental)
  Interventions: Drug: ARGX-113

INTERVENTIONS:
Drug: ARGX-113 — human IgG1-derived Fc fragment that binds to human neonatal Fc receptor (FcRn)

SUMMARY:
The proposed study is an open-label, non-controlled, adaptive-design Phase II study to evaluate the safety, pharmacodynamics, pharmacokinetics, efficacy, and conditions of use (dosage, frequency of administration at maintenance) of ARGX-113 in patients with mild to moderate Pemphigus (Vulgaris or Foliaceus), either newly diagnosed or relapsing.

The total study duration for each patient is less than 6 months. It consists of a Screening period, an Induction, a maintenance treatment period followed by a treatment-free Follow-up (FU) period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥ 18 years.
2. Clinical diagnosis of PV or PF, that has been confirmed by positive direct immunofluorescence and by positive indirect immunofluorescence and/or ELISA.
3. Mild to moderate disease severity (PDAI < 45).
4. Newly diagnosed patients or relapsing patients off therapy with or without a first course of prednisone of maximum 4 weeks, and for whom an initial period of ARGX-113 monotherapy is judged clinically acceptable; or newly diagnosed patients or relapsing patients off therapy on a first course of oral prednisone at stable dose for at least 2 weeks and for whom ARGX-113 monotherapy is considered not clinically acceptable; or patients who relapse despite oral prednisone at tapered dose +/- a conventional immunosuppressant (e.g. azathioprine, mycophenolate mofetil).
5. Identified serum levels of autoantibodies directed against Dsg 3 and/or Dsg-1 antigens at screening, using indirect immunofluorescence or ELISA.
6. Ability to understand the requirements of the study, provide written informed consent (including consent for the use and disclosure of research-related health information), and comply with the study protocol procedures (including required study visits).

Exclusion Criteria:

1. Pregnant and lactating women, and those intending to become pregnant during the study or within 90 days after the last dosing. Women of childbearing potential should have a negative serum pregnancy test at Screening and a negative urine pregnancy test at Baseline, prior to administration of IMP.
2. Male patients who are sexually active that do not intend to use effective methods of contraception during the study or within 90 days after the last dosing.
3. Confirmed diagnosis of paraneoplastic pemphigus, drug-induced pemphigus or any other non-PV/non-PF autoimmune blistering disease.
4. History of refractory disease to active third line therapy (e.g. intravenous polyvalent human immunoglobulins [IVIg], rituximab, plasma exchange/ immunoadsorption).
5. Use of therapies other than oral prednisone and conventional immunosuppressants, that can interfere in the clinical course of the disease (e.g. intravenous [IV] prednisolone bolus, dapsone, sulfasalazine, tetracyclines, nicotinamide, plasmapheresis/ plasma exchange, immunoadsorption and IVIg) within 2 months prior to Baseline visit.
6. Use of rituximab and other CD20 target biologics within 6 months prior to Baseline visit.
7. History of anaphylactic reaction, or a known hypersensitivity reaction to one of the components of the IMP.
8. History of vaccination within the last 4 weeks prior to Baseline visit, or with a planned vaccination during the study, with the exception of seasonal vaccination (e.g. influenza vaccine).
9. Recent serious infection (i.e., requiring injectable antimicrobial therapy or hospitalization) within the 8 weeks prior to Baseline visit.
10. Known active or chronic viral infection with hepatitis B virus (HBV); refer to the Centers for Disease Control and Prevention (CDC) guidelines.
11. Known seropositive or active infection with hepatitis C virus (HCV).
12. Known history of or known viral infection with human immunodeficiency virus (HIV 1 and 2 antibodies).
13. Body Mass Index (BMI) at Screening > 35,0 kg/m2.
14. Clinical evidence of significant active, unstable or uncontrolled concomitant disease (e.g. cardiovascular, pulmonary, hematologic, gastrointestinal, endocrinological and metabolic, hepatic, renal, neurologic, malignancy, infectious diseases, coagulopathies, other autoimmune disease) or condition (lack of peripheral venous access, recent major surgery, etc), which, in the opinion of the investigator, puts the patient at undue risk or may affect the interpretation of the results.
15. Patients in general health condition not allowing study participation (Karnofsky index < 60%; see Appendix 14.2).
16. At Screening, have clinically significant laboratory abnormalities as below:

    1. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 × upper limit of normal (ULN)
    2. Total serum bilirubin of > 1.5 x ULN (except for Grade 1 hyperbilirubinemia as defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), due solely to a documented medical diagnosis of Gilbert's syndrome)
    3. Serum creatinine of > 1.5 mg/dL or creatinine clearance < 50 mL/min (using the Chronic Kidney Disease Epidemiology Creatinine formula)
    4. Hemoglobin (Hb) ≤ 9 g/dL
    5. International normalized ratio (INR) > 1.5 or activated partial thromboplastin time (aPTT) > 1.5 x ULN
    6. Total immunoglobulin G (IgG) level < 6 g/L
    7. Presence of > 1 + proteinuria dipstick
17. Patient having participated in another interventional study within the last 3 months prior to Baseline visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2020-10-28 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as measured by the incidence and severity of treatment-emergent (serious) adverse events over the study. | Up to 6 months

SECONDARY OUTCOMES:
Evaluation of serum levels of total IgG and subtypes (IgG1, IgG2, IgG3, IgG4) | Up to 6 months
Evaluation of serum levels of anti Dsg-1 and -3 autoantibodies | Up to 6 months
Pemphigus Disease Area Index (PDAI) | Up to 6 months
  The score has a range from 0 to 263, the higher the score, the more severe the disease.
Time to disease control (DC), control being defined as the absence of new lesions and established lesions beginning to heal | Up to 6 months
Time until relapse, relapse being defined as the appearance of 3 or more new lesions a month that do not heal spontaneously within 1 week, or as the extension of established lesions | Up to 6 months
Pharmacokinetic parameters of ARGX 113: Tmax | Up to 6 months
Pharmacokinetic parameters of ARGX 113: Cmax | Up to 6 months
Incidence of anti-drug antibodies (ADA) to ARGX 113 | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Dupuy, MD, Study Director — argenx
Locations (12):
- Germany (2):
  - University of Lübeck and UKSH, Department of Dermatology and Lübeck Institute of Experimental Dermatology, Lübeck
  - Clinic of Dermatology and Allergology - Philipps University Marburg, Marburg
- Hungary (3):
  - University of Debrecen Medical Center Department of Dermatology, Debrecen
  - University of Pécs Clinical Center , Department of Dermatology, Venerology and Oncodermatology, Pécs
  - University of Szeged Faculty of Medicine Albert Szent-Györgyi Medical Center Department of Dermatology and Allergology, Szeged
- Israel (3):
  - HaEmek Medical center, Dermatology Department, Afula
  - Department of Dermatology, The Chaim Sheba Medical Center, Tel Aviv
  - Department of dermatology, The Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (2):
  - Dermopathic Institute of the Immaculate - Foundation "Luigi Maria Monti", Rome
  - Foundation Policlinico A. Gemelli - Dermatology Department, Rome
- Ukraine (2):
  - National Medical University named after O.O.Bohomolets, Department of Dermatology and Venereology based on Oleksandrivska Clinical Hospital of Kyiv City, Department of Dermatology, Kyiv
  - Municipal Institution "Zaporizhzhya Regional Dermatology and Venereology Clinical Dispensary" of Zaporizhzhya Regional Council, Zaporizhzhya

REFERENCES:
- [Derived] Maho-Vaillant M, Sips M, Golinski ML, Vidarsson G, Goebeler M, Stoevesandt J, Bata-Csorgo Z, Balbino B, Verheesen P, Joly P, Hertl M, Calbo S. FcRn Antagonism Leads to a Decrease of Desmoglein-Specific B Cells: Secondary Analysis of a Phase 2 Study of Efgartigimod in Pemphigus Vulgaris and Pemphigus Foliaceus. Front Immunol. 2022 May 18;13:863095. doi: 10.3389/fimmu.2022.863095. eCollection 2022. PMID 35663943
- [Derived] Goebeler M, Bata-Csorgo Z, De Simone C, Didona B, Remenyik E, Reznichenko N, Stoevesandt J, Ward ES, Parys W, de Haard H, Dupuy P, Verheesen P, Schmidt E, Joly P; ARGX-113-1701 Investigator Study Group. Treatment of pemphigus vulgaris and foliaceus with efgartigimod, a neonatal Fc receptor inhibitor: a phase II multicentre, open-label feasibility trial. Br J Dermatol. 2022 Mar;186(3):429-439. doi: 10.1111/bjd.20782. Epub 2021 Nov 28. PMID 34608631